CLINICAL TRIAL: NCT00863824
Title: Elimination of NNAL and Cotinine From Hair and Urine
Brief Title: Clearance of NNAL and Cotinine From Second-hand Smoke in Hair and Urine
Acronym: NNAL
Status: Withdrawn | Type: Observational
Why Stopped: Study was not funded
Sponsor: University of Nebraska (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 0121-09-EP
Record Dates: First submitted 2009-03-17; First posted 2009-03-18 (Estimated); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Lung Cancer
Keywords: NNAL; Cotinine; Second hand smoke
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study will investigate how long it takes for NNAL and cotinine, markers of second hand smoke, to clear the human body.

DETAILED DESCRIPTION:
The purpose of the study is to investigate how long it takes for NNAL and cotinine, both specific markers of second hand tobacco smoke exposure to clear the human body.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Caucasians and African-Americans 19 years of age or above, how are ready to quit smoking

Exclusion Criteria:

* Anyone who is not a Caucasian or an African-American, below 19 years of age, and is currently taken prescription medication.

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Caucasians and African Americans who are ready to quit smoking.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-07 (Estimated); Primary Completion 2010-05-11 (Actual); Study Completion 2010-05-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chandran Achuatn, PhD, Principal Investigator — University of Nebraska